CLINICAL TRIAL: NCT07340580
Title: Facilitating Health System Implementation of Physical Activity Screening and Referral to Community-Based Programs: Exercise is Medicine Greenville
Brief Title: Implementation Facilitation of Exercise is Medicine Greenville
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: University of South Carolina School of Medicine, Greenville (Unknown); University of Nebraska (Other); University of Utah (Other); Temple University (Other); Prisma Health-Upstate (Other); Durham University (Other)
Responsible Party: Principal Investigator, Jennifer Trilk, Professor of Biomedical Sciences, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01HL173601-01A1 (NIH)
Record Dates: First submitted 2026-01-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Physical Inactivity; Dyslipidemia; Obesity and Overweight; Hypertension; Diabetes; Health Care Delivery; Patients; Chronic Disease; Exercise; Physical Activity; Implementation Science
Keywords: Implementation Facilitation; Physical activity referral scheme; Effectiveness-implementation hybrid type 3; Pragmatic design; Stepped wedge
MeSH Terms: conditions — Sedentary Behavior; Dyslipidemias; Obesity; Overweight; Hypertension; Diabetes Mellitus; Chronic Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will utilize a pragmatic, stepped wedge, cluster randomized design to examine the impact of implementation facilitation (IF) on increasing the reach (eligible patients that receive an EIMG referral) at 35 Prisma Health primary care clinics where the EIMG model is currently activated.
  At six-month intervals, randomly selected clinics will receive IF. We will use a mixed methods approach to explore factors related to achieving optimal implementation and reach of EIMG. We also will explore patient enrollment, participation, and dose-response relationships associated with changes in PA levels, health outcomes, and cost savings to the health system. Throughout the study, we will identify successful IF strategies across clinic settings, helping us identify and address potential inequities in the types of patients who receive EIMG referrals, are engaged in the EIMG referral pathway, and enroll and complete the community-based PA program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinic Implementation Facilitation (Experimental): Clinics will work with the facilitation team to address barriers and improve clinic workflow to increase patient referral rates to the community PA program.
  Interventions: Behavioral: Clinic Implementation Facilitation

INTERVENTIONS:
Behavioral: Clinic Implementation Facilitation — This single arm intervention will be applied to 35 Prisma Health primary care clinics where the EIMG model is currently activated. At six-month intervals, six or more clinics will receive tailored implementation facilitation (IF) based on pre-implementation facilitation findings at each clinic. We will explore factors related to achieving optimal implementation and reach of EIMG. Patient referral rates and health outcomes will also be captured as a result of changes of clinical workflow due to the IF.

SUMMARY:
A public health priority exists for the U.S. healthcare sector to integrate physical activity (PA) as a part of the patient care model. This research will provide valuable information on facilitating optimal implementation of a clinic-to-community model that identifies, refers, and enrolls physically inactive patients to community-based PA programs for the prevention and treatment of chronic diseases. Further, this work will provide evidence on the cost-effectiveness of integrating PA in healthcare systems as a population health management strategy.

DETAILED DESCRIPTION:
There is great potential for promoting physical activity (PA) for chronic disease prevention and treatment through the health care sector. Research has demonstrated effectiveness in assessing patient PA levels, providing 'exercise prescriptions', and referring patients to evidence-based PA programs in community settings. However, implementation barriers exist, ranging from practice integration to information flow, resulting in no major health systems integrating PA as part of a comprehensive approach to patient care. In 2016, a multi-organizational partnership between a large academic healthcare system, an academic institution, and a national PA organization launched Exercise is Medicine Greenville (EIMG), a comprehensive clinic-to-community approach that involves PA assessment, prescription, and referral of patients with chronic diseases to a tailored, community-based PA program. Since 2016, EIMG has expanded to 35 Prisma Health primary care clinics and 7 community PA facilities covering >400 square miles. Despite referring >1900 patients to date, great variability exists across participating clinics in correctly identifying eligible patients and providing EIMG referrals, reducing the overall reach and efficiency of engaging patients in the community-based PA programs. Using a pragmatic, stepped wedge, cluster randomized design, this research will examine the impact of implementation facilitation (IF) on improving the implementation and reach of EIMG with patients visiting participating Prisma Health primary care clinics. At six-month intervals, 35 randomly selected clinics (6 clinics in wave 1, 8 clinics in wave 2, 10 clinics in wave 3, and 11 clinics in wave 4) will receive IF planning (3 months), active IF (6 months), and post-IF maintenance (min 12 months). The specific aims of this project are to: 1) determine differences in the level of implementation (i.e., delivery fidelity) and reach (i.e., number, proportion, representativeness of patients) at Prisma primary care health clinics before and after IF, 2) assess levels of patient engagement in and the effectiveness of the 12-week, community-based PA programs, and 3) evaluate the costs of IF and the effects of increased EIMG referrals to the community-based PA program on patients costs and clinical outcomes. The mixed methods evaluation approach is guided by the RE-AIM framework to inform the assessment of implementation outcomes, and the i-PARIHS framework to describe contextual factors (i.e., determinants) influencing patient and clinic level outcomes. Through this work, the research will identify successful IF strategies across heterogeneous health settings, helping to identify and address potential inequities in the types of patients that receive EIMG referrals, are engaged in the EIMG referral pathway, and enroll and complete the community-based PA program. Study findings will provide important information on improving future implementation and scalability of PA integration in large health systems, optimizing clinic-community linkages, and the cost savings related to primary and secondary prevention of cardiovascular disease-related health outcomes in the general patient population.

ELIGIBILITY:
The primary aim of this study is implementation facilitation at the clinic level. The secondary aim of this study is at the patient level. Therefore we have divided our inclusion/exclusion eligibility criteria by primary and secondary aim.

1. Clinic (primary aim) Inclusion criteria

* Currently EIMG-activated Prisma Health-Upstate Primary Care clinics (family or internal medicine)
* Adopted EIMG >= 6 months prior to the beginning of this study

  1. Clinic (primary aim) Exclusion criteria
* Not EIMG-activated
* Adopted EIMG < 6 months prior to the beginning of this study
* Greater than 15 miles from the nearest YMCA

  1. Primary care clinic staff (primary aim) Inclusion criteria
* At least 18 years of age
* Worked at the Prisma Health-Upstate clinic a minimum of three months
* Able to understand and communicate in English

  1. Primary care clinic staff (primary aim) Exclusion criteria
* Less than 18 years of age
* Worked at the Prisma Health-Upstate clinic less than three months
* Unable to speak or understand English
* Adults unable to provide consent

  2. Patient (secondary aim) Inclusion criteria (must meet all of below)
* Age >= 18 and <= 80 years
* Clinically eligible (diagnosis of hypertension, dyslipidemia, obesity, diabetes, or physical inactivity) to receive an EIMG referral
* A healthcare visit with an eligible encounter type (evaluation, telemedicine, consult, office visit, e-visit, follow-up, appointment, education, multidisciplinary visit, nutrition, occupational medicine-office visit)
* A healthcare visit at a participating clinic

  2. Patient (secondary aim) Exclusion criteria
* Age < 18 or > 80 years
* Current referral to Physical therapy or occupational therapy
* Current referral to cardiac, pulmonary, or oncology rehab
* One of the following visit diagnoses listed below:

  * Alzheimer's disease
  * Amyotrophic lateral sclerosis
  * angina or chest pain
  * congenital stenosis of aortic valve
  * congenital insufficiency of aortic valve
  * moderate or severe persistent asthma
  * typical or atypical atrial flutter
  * autonomic dysreflexia
  * acute bronchitis
  * cerebral infarction
  * encounter for chemotherapy
  * chronic kidney disease (stage 3-5)
  * end stage renal disease
  * coma
  * acute chronic obstructive pulmonary disease
  * unspecified dementia
  * dependence on renal dialysis
  * trisomy 21
  * pulmonary embolism
  * venous embolism and thrombosis
  * history of falling
  * acute fracture
  * left ventricular failure
  * congestive heart failure
  * hypertensive urgency, emergency or crisis
  * diabetes with ketoacidosis
  * chronic respiratory failure
  * dependence on supplemental oxygen
  * myocardial infarction
  * osteoporosis with current fracture
  * encounter for palliative care
  * paraplegia or quadriplegia
  * Parkinson disease
  * pneumonia
  * encounter for supervision of pregnancy
  * encounter for radiation therapy
  * serious mental illness (schizophrenia, psychotic disorder)
  * homicidal or suicidal ideations
  * sepsis
  * injury of spinal cord
  * presence of coronary stent
  * dependence on wheelchair or ambulatory aid

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinic-level differences in implementation of EIMG and reach of patients receiving EIMG referrals pre- and post-implementation facilitation | From Wave 1 start in pre-implementation facilitation activities to the end of Wave 4 post-implementation facilitation. Time frame for Wave 1 = 39 months, Wave 2 = 33 months, Wave 3 = 27 months, Wave 4 = 21 months.
  Reach (primary study outcome measure) will be assessed by estimating the number and proportion of eligible patient visits engaged in EIMG by providers. A patient's visit will be considered 'engaged' if they receive an EIMG referral. The proportion is estimated by dividing patient visits with an EIMG referral by all eligible patient visits. Reach will be calculated by provider and aggregated at the clinic level.
  Adoption will be assessed at the provider level by determining the number, proportion, and representativeness (i.e., sex, age, specialty) of providers that utilize any EIMG component in their practice compared to peers that do not use EIMG.
  Implementation will be assessed by determining the extent to which all three steps of EIMG (i.e., assessment, prescription, patient referral) are conducted with each eligible patient at the provider level, aggregated at the clinic level.

SECONDARY OUTCOMES:
Effectiveness of participating in the community-based, 12-week evidence-informed PA program on patient PA levels and health outcomes | From the time the patient is referred to the PA program to 12 months after the patient graduates from the program
  Effectiveness is the degree to which participating in the evidence-informed PA programs improves patient PA levels and health outcomes (i.e., changes in cardiometabolic biometric values).
  Patient PA levels will be evaluated using the PAVS and objective measurement (accelerometry) before starting the PA program, after completion of the PA program, and 12 weeks post-PA program.
  Patient health outcomes (i.e., body weight, blood pressure, hemoglobin A1c, lipid profiles) will be extracted from the Prisma Health electronic health record (EHR) at time of referral, after completion of the PA program, and at least 12 months after the PA program.
Cost of implementation facilitation and to estimate the effectiveness of increased EIMG referrals to the community-based PA on patient costs | IF costs will be measured from start of the Pre-IF phase to end of the IF phase (9 months) for each wave. For episode specific cost, measurements are taken from the index visit (day 0) within each episode through the end of the episode of care (day 240)
  Each ambulatory visit with an EIMG eligible diagnosis will serve as the standard unit of observation. Episodes of care will be defined after each visit through the end of follow-up and cost information will be summarized across each episode of care. For each episode of care we will extract from the EHR all healthcare utilization that occurred during the episode by type and quantity. Utilization types during the episode will be designated by Healthcare Common Procedure Coding System (HCPCS), Diagnosis Related Group (DRG), and National Drug (NDC) codes. In addition, we will use the REDCap-based data file to measure implementation costs and capture activity during the 12-week PA program. To obtain standardized costs across episodes, we will apply Prisma standard resource unit prices to all healthcare utilization. For each visit episode we will calculate Episode Healthcare Costs as the price-weighted sum of all healthcare resources used by patient "i" during the episode of care.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Trilk, PhD, Principal Investigator — University of South Carolina School of Medicine, Greenville
Locations (1):
- Prisma Health - Upstate, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided